CLINICAL TRIAL: NCT00258700
Title: Demonstrate Non-inferiority of Men-C Immune Response of Hib-MenC With Infanrix™-IPV Versus a Licensed Men-C Vaccine With Pediacel™ When Given at 2, 3, 4 Months and the Immunogenicity of Hib-MenC When Given as a Booster Dose at 12-15 Months
Brief Title: Primary & Booster Immunogenicity Study of GSK Biologicals' Hib-MenC Versus a Licensed Men-C Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 103974 (primary study); 104056 (Other: GSK)
Record Dates: First submitted 2005-11-24; First posted 2005-11-28 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines

INTERVENTIONS:
Biological: Haemophilus influenzae type b- and meningococcal (vaccine)

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of the candidate Hib-MenC conjugate vaccine co-administered with Infanrix™-IPV versus a licensed meningococcal serogroup C vaccine co-administered with Pediacel™ when given according to a 2, 3, 4 month schedule and the immunogenicity of the Hib-MenC vaccine when given as a booster dose at 12-15 months of age.

DETAILED DESCRIPTION:
This multicenter study is open with respect to the treatment allocation, but double-blind with respect to the Hib-MenC-TT lots (3 lots). The study will be conducted in two stages. Primary vaccination phase: 3 doses Hib-MenC-TT with Infanrix™-IPV or for the control group a licensed Men-C vaccine with Pediacel™ at 2, 3, 4 months of age; Booster/persistence phase: 1 dose Hib-MenC with Priorix™. 4 blood samples of 3.5ml (5ml for the UK subset) are collected (Study Months 0 & 3, prior to & 42 days after the booster).

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female, between, and including, 6 and 12 weeks of age.
* Born after a gestation period between 36 and 42 weeks
* Vaccination with hepatitis B at birth and at 6 to 12 weeks (concomitantly with the first study vaccine), accepted although not mandatory

Exclusion criteria:

* Planned administration/ administration of a vaccine not foreseen by the study protocol since birth, with the exception of Bacille Calmette Guerin (BCG) and hepatitis B vaccines.
* History of H. influenzae type b and /or meningococcal serogroup C disease.
* Previous vaccination against meningococcal serogroup C disease, diphtheria, tetanus, pertussis, polio or Hib disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* A family history of congenital or hereditary immunodeficiency
* History of any neurologic disorders or seizures
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 478 (Actual)
Dates: Start 2005-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
1 m after the 3rd dose of primary vaccination: SBA-MenC titre ≥ 1:8 (seroprotection status), anti-PRP concentration ≥ 0.15 µg/ml. 42 d after the booster vaccination: SBA-MenC titre ≥ 1:128, anti-PRP concentration ≥ 1 μg/ml

SECONDARY OUTCOMES:
Antibody levels to all vaccine antigens:1 m post dose 3, prior to & 42 d post booster. After each dose: Solicited (d 0-3, local & general), unsolicited (d 0-30) & MMR specific (d 0-42) symptoms. SAEs (whole study).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Poland (9):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Łęczna
- GSK Investigational Site, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pace D, Snape M, Westcar S, Oluwalana C, Yu LM, Begg N, Wysocki J, Czajka H, Maechler G, Boutriau D, Pollard AJ. A novel combined Hib-MenC-TT glycoconjugate vaccine as a booster dose for toddlers: a phase 3 open randomised controlled trial. Arch Dis Child. 2008 Nov;93(11):963-70. doi: 10.1136/adc.2007.136036. Epub 2008 May 7. PMID 18463125
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 103974 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103974 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103974 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103974 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103974 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 103974 (primary study) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register